CLINICAL TRIAL: NCT05916053
Title: Association Between Three-Months Vitamin D Supplementation and Depressive Symptomatology Incidence Among Saudi Arabian Adults
Brief Title: Supplementation and Depressive Symptomatology Incidence Among Saudi Arabian Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lebanese American University (Other)
Responsible Party: Principal Investigator, Rashel S. Khaddaj, Principal Investigator, Lebanese American University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LAU.SAS.BR2.12/Sep/2021
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Vitamin D Deficiency; Depressive Symptoms
MeSH Terms: conditions — Vitamin D Deficiency; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Nutritional education about food sources of vitamin D
- VItamin D supplemented (Experimental): Vitamin D supplementation of 50.000 IU weekly for 3 months.
  Interventions: Dietary Supplement: Vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation — 50.000 IU of vitamin D supplementation was prescribed for deficient/insufficient participants for a 3 month period.
  Arms: VItamin D supplemented

SUMMARY:
The goal of this randomized controlled trial is to explore the relationship between Vitamin D supplementation and depressive symptomatology in Saudi Arabian Population.

The main questions it aims to answer are:

* Is Vitamin D deficiency associated with an increased prevalence of depressive symptomatology among Saudi Arabian Population?
* Is Vitamin D Supplementation for a period of 3-month at 50,000 International Units might be associated with an improved depressive status? All the participants were clients who attended the clinic to help with weight management - who were doing regular medical check-ups - at Al Themal Medical Center which is located in Abha, Saudi Arabia.

Participants were requested to do a general blood test to check for any vitamins and minerals deficiencies as part of the routine clinical procedure. This procedure did not incur any additional costs on the behalf of the participants. The participants who were identified to have any deficiencies were recommended to take supplements, also as part of the routine clinical procedure. Therefore, participants identified to be deficient or insufficient Vitamin D levels were screened and recruited to participate in the current study.

Participants were randomly assigned to either an interventional (vitamin D) or placebo group (control). The interventional group received vitamin D supplementation of 50.000International Units/week for 3 months and the placebo group received dietary advice and education on food sources of vitamin D for the same period. Both Groups received a weight gain or a weight loss diet as per their case.

At the three-months follow-up, the participants were readministered the face-to-face questionnaire and their blood levels for vitamin D were also checked.

Thus, this study would add value to the actions taken to treat vitamin D deficiency in Saudi Arabian adults. This might also assist in approaching new recommendations related to preventing or treating depression via vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females Aged between 18 and 65 years old
* Be Vitamin D deficient/Insufficient (As tested via blood levels)
* Have a BMI between 17kg/m2 & 55 kg/m2
* Able to understand Arabic
* Able to provide written consent

Exclusion Criteria:

* Participants already taking Vitamin D supplements or Anti-depressants
* Participants having normal vitamin D levels
* Participants reporting other mental health diseases
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptomatology | 3 months supplementation
  Assess depressive symptomatology via Patient Health Questionnaire-9. The lower the score, the better the outcome. The scores of the Patient Health Questionnaire-9 were interpreted as follows: 0-4 Minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Rahi, PHD, Study Director — Sam Houston State University
Locations (1):
- Al Themal Medical Center, Abhā, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No